CLINICAL TRIAL: NCT05997147
Title: Development and Validation of a Preoperative Model to Predict the Lymphovascular Invasion of Pancreatic Ductal Adenocarcinoma: a Multicenter Retrospective Study
Brief Title: A Preoperative Model to Predict the Lymphovascular Invasion in Pancreatic Ductal Adenocarcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Panc-LVI-2023810
Record Dates: First submitted 2023-08-10; First posted 2023-08-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Predictive Cancer Model; Pancreas Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Importance: Lymphovascular invasion (LVI) is a poor prognosis pathologic feature in pancreatic ductal adenocarcinoma (PDAC) patients. Neoadjuvant therapy may bring survival benefits to these patients.

Objective: To construct a preoperative model which could predict LVI in PDAC patients and further validate it in other cohorts.

Design, Setting, and Participants: Patients from 3 three tertiary hospitals were included in this study. Univariate and multivariate Logistic regression analyses were conducted to define independent prediction factors of LVI. A nomogram was constructed based on the result of multivariate analysis.The predictive value of the model was assessed using receiver operating characteristic (ROC) curves and the maximum Youden index of the ROC curve was defined as the cut-off point. The calibration plot was utilized to assess the concordance of the model. The decision curve analyses (DCA) were applied to estimate the clinical benefit of using this model to predict LVI.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were pathologically diagnosed as PDAC and received curative surgery.

Exclusion Criteria:

* Patients with distant metastasis; Patients who received neoadjuvant therapy; Patients with a survival time of less than 1 month.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were pathologically diagnosed as PDAC and received curative surgery.
Sampling Method: Non-Probability Sample
Enrollment: 1009 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-08-05 (Actual); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival | 10 years
  Time from operation to the detection of recurrence or last follow-up

SECONDARY OUTCOMES:
Overall survival | 10 years
  Time between surgical resection to death or the last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Jihui Hao, Dr, Study Chair — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China